CLINICAL TRIAL: NCT04919629
Title: Randomized Phase 2 Trial of APL-2 With Pembrolizumab vs. APL-2 With Pembrolizumab and Bevacizumab vs. Bevacizumab Alone in Patients With Recurrent Ovarian Cancer and Persistent Malignant Effusion
Brief Title: APL-2 and Pembrolizumab Versus APL-2, Pembrolizumab and Bevacizumab Versus Bevacizumab Alone for the Treatment of Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer and Malignant Effusion
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 798120; NCI-2021-04265 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 798120 (Other: Roswell Park Cancer Institute); R01CA267690 (NIH)
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Fallopian Tube Carcinosarcoma; Fallopian Tube Clear Cell Adenocarcinoma; Fallopian Tube Endometrioid Adenocarcinoma; Fallopian Tube Serous Adenocarcinoma; Ovarian Carcinosarcoma; Ovarian Clear Cell Adenocarcinoma; Ovarian Endometrioid Adenocarcinoma; Ovarian Serous Adenocarcinoma; Primary Peritoneal Carcinosarcoma; Primary Peritoneal Clear Cell Adenocarcinoma; Primary Peritoneal Endometrioid Adenocarcinoma; Primary Peritoneal Serous Adenocarcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; pegcetacoplan; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 2A-1 (pegcetacoplan, pembrolizumab) (Experimental): Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Patients also receive pembrolizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive pembrolizumab for up to 35 21-day cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Pegcetacoplan; Biological: Pembrolizumab; Other: Questionnaire Administration
- Cohort 2A-2 (pegcetacoplan, pembrolizumab, bevacizumab) (Experimental): Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Patients also receive pembrolizumab IV and bevacizumab IV on day 1of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive pembrolizumab for up to 35 21-day cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Pegcetacoplan; Biological: Pembrolizumab; Other: Questionnaire Administration
- Cohort 2B-1 (pegcetacoplan, pembrolizumab) (Experimental): (Expansion) Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV on day 1 of each cycle. Treatment repeats every 21 days for 6 cycles, followed by every 42 days for up to 35 total cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.
  Interventions: Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Pegcetacoplan; Biological: Pembrolizumab; Other: Questionnaire Administration
- Cohort 2B-2 (pegcetacoplan, pembrolizumab, bevacizumab) (Experimental): Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Patients also receive pembrolizumab IV and bevacizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive pembrolizumab for up to 35 21-day cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Pegcetacoplan; Biological: Pembrolizumab; Other: Questionnaire Administration
- Cohort 2B-3 (bevacizumab) (Experimental): Patients receive bevacizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.
  Interventions: Biological: Bevacizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Other: Questionnaire Administration

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; CT-P16; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Cohort 2A-2 (pegcetacoplan, pembrolizumab, bevacizumab); Cohort 2B-2 (pegcetacoplan, pembrolizumab, bevacizumab); Cohort 2B-3 (bevacizumab)
Procedure: Biopsy — Undergo tumor biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Pegcetacoplan — Given IV and SC
  Arms: Cohort 2A-1 (pegcetacoplan, pembrolizumab); Cohort 2A-2 (pegcetacoplan, pembrolizumab, bevacizumab); Cohort 2B-1 (pegcetacoplan, pembrolizumab); Cohort 2B-2 (pegcetacoplan, pembrolizumab, bevacizumab)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; Keytruda; Lambrolizumab; MK-3475; Pembrolizumab Biosimilar BCD-201; SCH 900475
  Arms: Cohort 2A-1 (pegcetacoplan, pembrolizumab); Cohort 2A-2 (pegcetacoplan, pembrolizumab, bevacizumab); Cohort 2B-1 (pegcetacoplan, pembrolizumab); Cohort 2B-2 (pegcetacoplan, pembrolizumab, bevacizumab)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the effect of APL-2 when given in combination with either pembrolizumab or pembrolizumab and bevacizumab compared with bevacizumab alone in treating patients with ovarian, fallopian tube, or primary peritoneal cancer that has come back (recurrent) and a buildup of fluid and cancer cells (malignant effusion). APL-2 may limit tumor progression, decrease malignant effusion production, and improve the immune system's response against cancer cells. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is a monoclonal antibody that may interfere with the ability of tumor cells to grow and spread. Giving APL-2 together with either pembrolizumab or pembrolizumab and bevacizumab may work better in treating patients with ovarian, fallopian tube, or primary peritoneal cancer and malignant effusion compared to bevacizumab alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety of pegcetacoplan (APL-2) alone and in combination with pembrolizumab, and APL-2 in combination with both bevacizumab and pembrolizumab in patients with recurrent ovarian cancer with symptomatic malignant effusion (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0).

II. Effect of therapy on of malignant effusion measured by total volume of effusion drained every 3 weeks (patient diary and/or drained volume).

SECONDARY OBJECTIVES:

I. Determine progression-free survival (PFS), objective response rate (ORR), disease control rate (DCR) and overall survival (OS) per immune related response criteria (irRECIST).

II. Changes in quality of life measures during the clinical trial (European Organisation for the Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire [QLQ]-Core 30 [C30], EORTC QLQ-Ovarian version 28 [OV28] and Multidimensional Fatigue Symptom Inventory-Short Form [MFSI-SF]).

EXPLORATORY OBJECTIVES:

I. Evaluate the immunologic and phenotypic changes in malignant effusions and blood samples in all cohorts, which can include the following:

Ia. To understand the signaling mechanisms in ascites primed neutrophils and their effects on tumor cell growth.

Ib. To understand the changes in complement activation pathways. Ic. Functional assays of neutrophil, macrophage and T cells. Id. Flow cytometry for immune cell composition. Ie. Luminex assay for circulation inflammatory cytokines/chemokines, angiogenesis markers.

II. In patients with solid tumor lesions accessible by image-guided core biopsies the effects of therapy will be determined on the immune composition of tumor microenvironment. Studies on tumor may include immune cell infiltration, ribonucleic acid (RNA)-sequencing (Seq) and T cell receptor (TCR)-Seq for immune cell activation and exhaustion markers, complement deposits, genomic and transcriptomic profile.

III. Microbiome analysis from stool, tumor tissue and malignant effusions. IV. Determine the concentration (pharmacokinetics [PK]/pharmacodynamics [PD]) of APL-2 in serum and malignant effusion.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP 2A: Patients are assigned to 1 of 2 cohorts.

COHORT 2A-1: Patients receive pegcetacoplan intravenously (IV) over 20-40 minutes on day 1 of cycle 1 and then subcutaneously (SC) twice weekly (BIW) of each cycle. Patients also receive pembrolizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive pembrolizumab for up to 35 21-day cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.

COHORT 2A-2: Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Patients also receive pembrolizumab IV and bevacizumab IV on day 1of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive pembrolizumab for up to 35 21-day cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.

GROUP 2B: Patients are assigned to 1 of 3 cohorts.

COHORT 2B-1: Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients also receive pembrolizumab IV on day 1 of each cycle. Treatment repeats every 21 days for 6 cycles, followed by every 42 days for up to 35 total cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.

COHORT 2B-2: Patients receive pegcetacoplan IV over 20-40 minutes on day 1 of cycle 1 and then SC BIW of each cycle. Patients also receive pembrolizumab IV and bevacizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients may receive pembrolizumab for up to 35 21-day cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.

COHORT 2B-3: Patients receive bevacizumab IV on day 1 of each cycle. Treatment repeats every 3 weeks for up to 7 cycles in the absence of disease progression or unacceptable toxicity. Patients undergo tumor biopsy and blood sample collection throughout the study.

After completion of study treatment, patients are followed up at 30 days and then every 12 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age on day of signing informed consent
* Recurrent epithelial ovarian/fallopian tube or primary peritoneal cancer (serous, clear cell, endometrioid, mixed or poorly differentiated or carcinosarcoma) based on imaging or synchronous primary ovarian and uterine cancer patients with any of the histology subtypes mentioned above regardless of platinum sensitivity, prior stage or number of prior treatment lines
* Symptomatic ascites or pleural effusion or both requiring >= 1 drainage within 4-weeks of study entry or has a peritoneal/pleural drainage catheter in place to control symptoms
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patient has not received pembrolizumab or other immune checkpoint inhibitor treatment for 9 weeks prior to enrollment
* Life expectancy of >= 3 months
* Absolute neutrophil count (ANC): >= 1,500/µL
* Platelets: >= 75,000/µL
* Hemoglobin: >= 9 g/dL or 5.6 mmol/L (within 7 days of assessment)
* Creatinine: =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance >= 60 mL/min (Cockcroft-Gault Equation) for participant with creatinine levels > 1.5 X institutional ULN. GFR can also be used in place of creatinine or creatinine clearance (CrCl)
* Total bilirubin: =< 1.5 X ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]): =< 2.5 X ULN OR =< 5 X ULN for participants with liver metastases
* Albumin: > 2.5 gm/dL
* International Normalized Ratio (INR) or Prothrombin Time (PT): =< 1.5 unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT): =< 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* A woman of childbearing potential must have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Participants of childbearing potential must be willing to use 2 methods of birth control or be surgically sterile or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication (participants of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year). Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately
* Willing and able to self-administer APL-2 (administration by caregiver will be allowed)
* No known absolute contraindication to bevacizumab and/or pembrolizumab treatment per enrolling provider
* Willing to receive vaccination against Neisseria meningitidis, Streptococcus pneumoniae, and Hemophilus influenzae if randomized into an APL-2 receiving arm, if not already vaccinated
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Is currently receiving any additional cancer therapy or participating or used an investigational drug or device within 3 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment or, is taking any other medication that might affect immune function
* Has active autoimmune disease that has required systemic treatment in the past 3 months (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Participant has clinically significant cardiovascular disease including:

  * Uncontrolled hypertension, defined as systolic >150 mmHg or diastolic >90 mmHg
  * Myocardial infarction or unstable angina within 6 months prior to enrollment
  * New York Heart Association (NYHA) Grade II or greater congestive heart failure
  * Participant has a Grade II (NYHA) or greater peripheral vascular disease
  * Participant has a clinically significant peripheral artery disease (e.g. those with claudication), within 6 months prior to study enrollment
* Pregnancy or lactation
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug
* Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Has a known history of human immunodeficiency virus (HIV) infection
* Concurrent active hepatitis B (defined as hepatitis B surface antigen [HBsAg] positive and/or detectable HBV deoxyribonucleic acid [DNA]) and hepatitis C virus (HCV) (defined as anti-HCV Ab positive and detectable HCV ribonucleic acid [RNA]) infection. Note: Hepatitis B and C screening tests are not required unless known history of HBV and HCV infection
* Has received any investigational vaccines (i.e., those not licensed or approved for emergency use). Note: Any licensed COVID-19 vaccine (including for Emergency Use) is allowed in the study as long as they are modified ribonucleic acid (mRNA) vaccines, adenoviral vaccines, or inactivated vaccines. These vaccines will be treated just as any other concomitant therapy. Investigational vaccines (i.e., those not licensed or approved for emergency use) are not allowed
* Known additional malignancy that is progressing or has required active treatment within the past 2 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (Phase 2a) | Up to 30 days after last dose
  Toxicities and adverse events (as per Common Terminology Criteria for Adverse Events version 5.0) will be summarized by cohort and grade using frequencies and relative frequencies.
Accumulation of effusion (Phase 2b) | Up to 3 years
  Will determine the effect of therapy on accumulation of effusion measured by total volume removed every 3 weeks. The change in accumulation of effusion (relative to pre-treatment) will be modeled as a function of cohort, time-point, their two-way interaction, baseline levels, and a random subject effect using a linear mixed model. The change will be compared: a) over-time within each cohort, and b) between the control cohort (cohort C) and each dosing cohort (cohorts A and B) using two-sided Bonferroni or Dunnet adjusted tests about the appropriate contrasts of model estimates. The model assumptions will be evaluated graphically, and transformations will be applied as appropriate.

SECONDARY OUTCOMES:
Overall survival | From treatment until death or last follow-up, assessed up to 3 years
  Will be summarized by cohort using standard Kaplan-Meier methods. As an exploratory analysis, the two dosing cohorts (cohorts A and B) may be compared to the control cohort (cohort C) compared using one-sided log-rank tests.
Progression free survival (PFS) | From treatment initiation until disease progression, death, or last disease assessment (censored), assessed up to 3 years
  Will be summarized by cohort using standard Kaplan-Meier methods, where estimates of median PFS are obtained with 90% confidence intervals. As an exploratory analysis, the two dosing cohorts (cohorts A and B) may be compared to the control cohort (cohort C) compared using one-sided log-rank tests.
Best response | Up to 3 years
  Will be summarized by cohort using frequencies and relative frequencies.
Overall response rate | Up to 3 years
  Defined as the proportion of patients who have a partial or complete response to therapy. Will be estimated by cohort using 95% confidence intervals obtained by Jeffrey's prior method.
Disease control rate | Up to 3 years
  Defined as the percentage of patients with advanced or metastatic cancer who have achieved complete response, partial response and stable disease. Will be estimated by cohort using 95% confidence intervals obtained by Jeffrey's prior method.
Quality of life (QOL) scores | Up to 3 years
  The QoL scores will be summarized by cohort and time-point using the appropriate descriptive statistics. Each QoL score will be model as a function of cohort, time, their two-way interaction, and a random subject effect using a linear mixed model. Comparisons between cohorts within timepoint or between timepoints within cohort will be made using tests about the appropriate contrasts of model estimates. All model assumptions will be evaluated graphically, and transformations will be applied as appropriate.

OTHER OUTCOMES:
APL-2 pharmacokinetics (PK)/pharmacodynamics (PD) and immunological | Baseline, day 1 of cycles 2, 3, and 7, and at end of treatment
  APL-2 measures and immune markers will be summarized by cohort and time-point using the appropriate descriptive statistics. Each measure will be model as a function of cohort, time, their two-way interaction, and a random subject effect using a linear mixed model. Comparisons between cohorts within timepoint or between timepoints within cohort will be made using tests about the appropriate contrasts of model estimates. All model assumptions will be evaluated graphically, and transformations will be applied as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Emese Zsiros, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States